CLINICAL TRIAL: NCT03802110
Title: Acute Feasibility Investigation of a New S-ICD Electrode Arrangement for Reduction of Defibrillation Energies
Brief Title: Acute Feasibility Investigation of a New S-ICD Electrode
Acronym: ASE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: C2081
Record Dates: First submitted 2018-11-08; First posted 2019-01-14 (Actual); Results first posted 2024-05-09 (Actual); Last update posted 2024-05-09 (Actual); Status verified 2023-10

CONDITIONS: Ventricular Fibrillation
MeSH Terms: conditions — Ventricular Fibrillation | interventions — Defibrillators, Implantable

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Single Arm (Experimental): Defibrillation threshold (DFT) testing Arm
  Interventions: Device: commercially released subcutaneous implantable cardioverter defibrillator (S-ICD) and the Investigational S-ICD Adapter.

INTERVENTIONS:
Device: commercially released subcutaneous implantable cardioverter defibrillator (S-ICD) and the Investigational S-ICD Adapter. — The S-ICD System is a Subcutaneous (under the skin) Implantable Cardioverter Defibrillator for people who are at risk of Sudden Cardiac Arrest. A new electrode configuration will be tested for Defibrillation testing ( DFT). The unit of measure will be in Joules. VF will be induced and the device will deliver a shock at a certain defined energy level as described in the protocol
  Other Names: The S-ICD System is a Subcutaneous (under the skin) Implantable Cardioverter Defibrillator for people who are at risk of Sudden Cardiac Arrest

SUMMARY:
This is an early-stage feasibility study. This study seeks to characterize the performance of the new electrode shock configuration with the S-ICD

DETAILED DESCRIPTION:
Background: The subcutaneous implantable cardioverter-defibrillator (S-ICD, EMBLEM®, Boston Scientific Corp) delivers 80 J shocks from an 8 cm left-parasternal coil (LPC) to a 59 cc left lateral pulse generator (PG). A system that defibrillates with lower energy could significantly reduce PG size. Computer modeling and animal studies suggest a 2nd shock coil either parallel (P) to LPC or transverse (T) from xiphoid to PG pocket would significantly reduce shock impedance and defibrillation threshold (DFT).

Objective: Acutely test defibrillation efficacy of P and T configurations in patients receiving an S-ICD.

Methods: Testing was performed in patients receiving a conventional S-ICD system (C) for standard indications. Patients at risk for conversion failure, stroke or infection were excluded. A 65 J success with the conventional S-ICD was required prior to investigational testing. A second electrode was temporarily inserted from the xiphoid incision using the same introducer and sheath tools and connected to the PG with an investigational Y-adapter (Model 3598, Boston Scientific). Phase 1 (n=11) tested only P at a starting energy of 50 J with subsequent tests at 65 or 30 J then 40 or 20 J depending upon outcome. Phase 2 (n=21) tested both P and T in random order, starting at 30 J then either 40 or 20 J.

ELIGIBILITY:
Key Inclusion Criteria:

1. Subject is scheduled to receive a de novo S-ICD system implant per labeled indication.
2. Passing S-ICD screening ECG performed per applicable user's manual.
3. Subject is willing and capable of providing informed consent specific to local and national laws.
4. Subject is age 18 or above, or of legal age to give informed consentspecific to local and national law.

Key Exclusion Criteria:

1. Subject has an unusual chest anatomy (eg. pectus excavatum and pectus carinatum) that might impede the ability to temporarily insert a second S-ICD electrode.
2. Subject has a left ventricular ejection fraction ≤ 20% within 3 months prior to enrollment.
3. Subject has NYHA Class IV or unstable Class III heart failure.
4. Subject that, in the opinion of the investigator, cannot tolerate the DFT testing required by this protocol.
5. Subject is morbidly obese, defined as BMI ≥ 35.
6. Subject has an active infection or has been treated for infection within the past 30 days.
7. Subject that, in the opinion of the investigator, has an increased risk of infection.
8. Subject is currently requiring/receiving dialysis.
9. Subject has insulin-dependent diabetes.
10. Subject had/has any prior or planned other surgical procedure within ±30 days of enrollment.
11. Subject that, in the opinion of the investigator, has an increased risk for thromboembolic event.
12. Subject that, in the opinion of the investigator, has an increased risk of excessive bleeding.
13. Subject is currently on an active heart transplant list.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2018-11-29 (Actual); Primary Completion 2022-04-01 (Actual); Study Completion 2022-04-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Reinoud Knops, Principal Investigator — Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Locations (4):
- Netherlands (4):
  - Academisch Medisch Centrum, Amsterdam
  - St. Antonius Ziekenhuis, Nieuwegein
  - Erasmus MC - University Medical Center Rotterdam, Rotterdam
  - Isala Klinieken, Zwolle

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects who were scheduled to receive an subcutaneous implantable cardioverter defibrillator (S-ICD), and fulfilled the inclusion and exclusion criteria, could be approached for enrollment and consent within 30 days of their scheduled implant.
Groups:
- Acute Test: Subjects who signed the Informed Consent Form (ICF) and were considered enrolled.
Period: Overall Study
Arm/Group | Acute Test
Started | 42
Started Testing | 35
Completed | 28
Not Completed | 14

BASELINE CHARACTERISTICS:
Population: 35 subjects began the S-ICD implant with the intention of perfroming acute investigational testing
Groups:
- Acute Test: Subjects receiving a commercial S-ICD system for per manufacturer indications and medical society guidelines
Arm/Group | Acute Test
Number analyzed (Participants) | 35
Age, Continuous [Mean (Standard Deviation); unit: years] | 51 (17)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 28
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Netherlands | 35
Left Ventricular Ejection Fraction [Mean (Standard Deviation); unit: percent] | 40 (15)

OUTCOME MEASURES:

1. Primary Outcome: Defibrillation Threshold (DFT) of the New Shock Electrode Configuration in Joules
Description: The primary objective of this acute feasibility study is to measure the DFT of the new shock electrode configuration with an S-ICD system. The unit of measure will be in Joules. Ventricular Fibrillation (VF) will be induced and the device will deliver a shock at a certain defined energy level as described in the protocol
Time Frame: Acute- During the implant procedure- up to 1 hour
Population: transverse testing was added in phase 2, so fewer subjects tested. Only subjects completing testing were analyzed
Measure: Mean (Standard Deviation); unit: Joules
Groups:
- Parallel Shock Configuration: Acute VF conversion test: shock delivered from two left parasternal coil electrodes inserted in parallel to a left lateral PG
- Transverse Shock Configuration: Acute VF conversion test: shock delivered from left parasternal coil Plus transverse coil (xiphoid towards PG) to left lateral PG
Arm/Group | Parallel Shock Configuration | Transverse Shock Configuration
Number analyzed (Participants) | 33 | 20
Joules | 27.0 (8.8) | 31.5 (9.3)

2. Secondary Outcome: Number of Participants With Successful Ventricular Fibrillation (VF) Conversion at 40 Joules
Description: The secondary objective is to assess the conversion success of the new electrode configuration to convert VF. VF will be induced and the device will deliver a shock at a certain defined energy level as described in the protocol
Time Frame: Acute- During the implant procedure- up to 1 hour
Population: Transverse was added in Phase 2 so fewer subjects tested.
Measure: Count of Participants; unit: Participants
Arm/Group | Parallel Shock Configuration | Transverse Shock Configuration
Number analyzed (Participants) | 33 | 20
Participants | 32 | 18

ADVERSE EVENTS:
Time Frame: Reporting of events occurred during the period the subject was considered to be enrolled in the study: from implant up to 3 months after implant.
Arm/Group | Single Arm
All-Cause Mortality (participants affected / at risk) | 0/42
Serious Adverse Events (participants affected / at risk) | 1/42
Other Adverse Events (participants affected / at risk) | 16/42
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Single Arm (N=42)
Ventricular Fibrilation (Cardiac disorders) | 1 (1) — Failed S-ICD shock, 5 external shocks needed to convert, after start but before investigational procedure
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Single Arm (N=42)
Adverse Reaction-Allergic reaction (General disorders) | 1 (1)
Patient condition non-cardiovascular other (General disorders) | 1 (1)
Inappropriate Tachy Therapy Noise (Non-Cardiac) (Product Issues) | 3 (3)
Post surgical wound discomfort PG site (<30d post implant) (Injury, poisoning and procedural complications) | 1 (1)
Incisional/superficial infection(<30 d post implant without explant) (Injury, poisoning and procedural complications) | 1 (1)
Inadvertent Arrhythmia (Injury, poisoning and procedural complications) | 4 (4)
Hematoma-PG pocket (<or+ 30d post implant) (Injury, poisoning and procedural complications) | 2 (2)
Hemodynamic Instability (Injury, poisoning and procedural complications) | 1 (1)
S-ICD System Procedure Related - OTHER (Injury, poisoning and procedural complications) | 1 (1)
Incisional/superficial infection(>30d post implant) (Injury, poisoning and procedural complications) | 1 (1)

LIMITATIONS AND CAVEATS:
The study excluded certain patients believed to have the potential for higher DFTs and greater risk for AE.2 subjects were not tested with either two-electrode configuration due to requirement that VF must first be successfully converted in the Single configuration with 65 J. The sample size was small,subjects may have characteristics that do not perfectly match S-ICD recipients. In this cohort of patients from the Netherlands, age younger and BMI somewhat lower than what might occur in the US

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-01-20): https://cdn.clinicaltrials.gov/large-docs/10/NCT03802110/Prot_SAP_000.pdf